CLINICAL TRIAL: NCT03104985
Title: New Combined Laser Therapy in Patients With Trophic Ulcers of Lower Extremities and Chronic Venous Insufficiency
Brief Title: LLLT of Trophic Ulcers of Lower Extremities and Chronic Venous Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center Matrix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLLT-trophic-ulcers-Tula
Record Dates: First submitted 2017-03-21; First posted 2017-04-07 (Actual); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-02

CONDITIONS: Trophic Ulcers; Chronic Venous Insufficiency
Keywords: Trophic ulcer; low level laser therapy; Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Conventional treatment only.
  * An elastic compression of lower extremities: elastic bandages or compression hosiery of class 2
  * Pharmacotherapy: Anavenol, Aescusan, Glyvenol; drugs of the Benzopyrone group, including Troxevasin and Venoruton. Trental, Aspirin and Ticlid (Ticlopidine). Nonsteroidal anti-inflammatory drugs (Nimesil, OKI), various ointments containing Heparin, corticosteroids, as well as nonsteroidal anti-inflammatory drugs. Antibiotic therapy.
  * Topical treatment: in the presence of purulent discharge (phase I of the wound healing process) - bandaging with antiseptic solutions (1% Iodopiron solution, 0.1% Chlorhexidine solution) and hydrophilic ointments (Levosin, Levomecol). In phases II and III - after ulcer cleansing the preparations based on Hyaluronic acid (Curiozin).
  Interventions: Other: Conventional therapy
- Conventional therapy and combined LLLT (Experimental): Conventional therapy and combined LLLT (LASMIK device) was performed. External exposure was conducted on the 1-4 affected area during one session for 2 minutes per zone in pulsed mode, light pulse duration - 100-130ns, wavelength - 635nm, by a matrix emitter consisting of eight laser diodes with a surface area of 8cm2, at a distance of up to 7cm, with pulsed power of 40W. ILBI was conducted in continuous mode with wavelength between 365-405nm (UV-spectrum) and 520-525nm (green spectrum) alternately, during 12 daily treatment sessions according to the scheme:
  1. - 365-405nm, power 1-2mW, exposure 2 min;
  2. - 520-525nm, 1-2mW, 5 min;
  3. - 365-405nm, 1-2mW, 2 min;
  4. - 520-525nm, 1-2mW, 5 min;
  5. - 365-405nm, 1-2mW, 2 min;
  6. - 520-525nm, 1-2mW, 5 min;
  7. - 365-405nm, 1-2mW, 2 min;
  8. - 520-525nm, 1-2mW, 5 min;
  9. - 365-405nm, 1-2mW, 2 min;
  10. - 520-525nm, 1-2mW, 5 min;
  11. - 365-405nm, 1-2mW, 2 min;
  12. - 520-525nm, 1-2mW, 5 min
  Interventions: Device: LASMIK; Other: Conventional therapy

INTERVENTIONS:
Device: LASMIK — the physiotherapeutic device LASMIK (Registration Certificate in Russia № RZN 2015/2687 dated 25.05.2015).
  Arms: Conventional therapy and combined LLLT
Other: Conventional therapy — * An elastic compression of lower extremities,
  * Pharmacotherapy,
  * Topical treatment

SUMMARY:
The aim of this study was to evaluate comparatively the efficiency of traditional treatment methods in patients with chronic venous diseases of C6 class, and a new combined low level laser therapy (LLLT) by LASMIK device.

The results of outpatient examination and treatment of patients with venous trophic ulcers, observed in the City Polyclinic of "Tula Municipal Clinical Hospital №2" were analyzed.

DETAILED DESCRIPTION:
During a longitudinal study, a group of patients was followed up in the period of complete or partial recovery. International classification of lower extremity chronic venous disorders СЕАР was used as a clinical classification of chronic venous insufficiency (CVI).

Depending on the applied treatment method, patients were divided into 2 groups:

1. (n=34) Conventional treatment
2. (n=34) Conventional treatment + combined LLLT, including external exposure with 635nm wavelength + intravenous laser blood illumination (ILBI) with 365-405nm (UV-spectrum) and 520-525nm (green spectrum) wavelength alternately, according to the special scheme

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* CVI Stage 6 (S6) in compliance with СЕАР

Exclusion Criteria:

* hemorrhagic syndrome,
* neoplastic syndrome,
* hyperthermic syndrome (fever, patient body temperature over 38°C),
* syndrome of systemic (cardiac, vascular, respiratory, renal and hepatic) and multiple organ failure (general severe illness),
* cachexic syndrome (severe general exhaustion),
* epileptic syndrome,
* hysterical syndrome,
* convulsive syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Moskvin, Principal Investigator — State Scientific Center of Laser Medicine, Russia, Moscow
Locations (1):
- Tula Municipal Clinical Hospital №2, Tula, Russia

REFERENCES:
- See also: Educational website with publications, scientific articles, training manuals, guidelines, books on LLLT. — http://www.lazmik.ru

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Treatment: * An elastic compression of lower extremities: elastic bandages or compression hosiery of class 2
  * Pharmacotherapy: Anavenol, Aescusan, Glyvenol; drugs of the Benzopyrone group, including Troxevasin and Venoruton. Trental, Aspirin and Ticlid (Ticlopidine). Nonsteroidal anti-inflammatory drugs (Nimesil, OKI), various ointments containing Heparin, corticosteroids, as well as nonsteroidal anti-inflammatory drugs. Antibiotic therapy.
  * Topical treatment: in the presence of purulent discharge (phase I of the wound healing process) - bandaging with antiseptic solutions (1% Iodopiron solution, 0.1% Chlorhexidine solution) and hydrophilic ointments (Levosin, Levomecol). In phases II and III - after ulcer cleansing the preparations based on Hyaluronic acid (Curiozin).
  Conventional therapy: - An elastic compression of lower extremities,
  * Pharmacotherapy,
  * Topical treatment
- Conventional Therapy and Combined LLLT: External exposure was conducted on the 1-4 affected area during one session for 2 minutes per zone in pulsed mode, light pulse duration - 100-130ns, wavelength - 635nm, by a matrix emitter consisting of eight laser diodes with a surface area of 8cm2, at a distance of up to 7cm, with pulsed power of 40W. ILBI was conducted in continuous mode with wavelength between 365-405nm (UV-spectrum) and 520-525nm (green spectrum) alternately, during 12 daily treatment sessions according to the scheme:
  1. - 365-405nm, power 1-2mW, exposure 2 min;
  2. - 520-525nm, 1-2mW, 5 min;
  3. - 365-405nm, 1-2mW, 2 min;
  4. - 520-525nm, 1-2mW, 5 min;
  5. - 365-405nm, 1-2mW, 2 min;
  6. - 520-525nm, 1-2mW, 5 min;
  7. - 365-405nm, 1-2mW, 2 min;
  8. - 520-525nm, 1-2mW, 5 min;
  9. - 365-405nm, 1-2mW, 2 min;
  10. - 520-525nm, 1-2mW, 5 min;
  11. - 365-405nm, 1-2mW, 2 min;
  12. - 520-525nm, 1-2mW, 5 min
Period: Overall Study
Arm/Group | Conventional Treatment | Conventional Therapy and Combined LLLT
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Conventional Treatment: Conventional treatment only.
- Conventional Therapy and Combined LLLT: Conventional therapy and combined LLLT (LASMIK device)
- Total: Total of all reporting groups
Arm/Group | Conventional Treatment | Conventional Therapy and Combined LLLT | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Full Range); unit: years] | 56.9 [39 to 77] | 57.5 [40 to 78] | 57.2 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Trophic Ulcer Healing
Description: Number of participants with ulcer epithelialization was counted in both groups. Trophic ulcer healing in 6 months occurred in larger number of participants of conventional therapy and combined LLLT group.
Time Frame: 6 months follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | Conventional Therapy and Combined LLLT
Number analyzed (Participants) | 34 | 34
Participants | 11 | 28

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Conventional Treatment | Conventional Therapy and Combined LLLT
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No